CLINICAL TRIAL: NCT07230210
Title: The Effectiveness of Smart Technology Interventions Combining Nutrition and Exercise for Older Adults at Risk of Sarcopenia
Brief Title: Smart Tech-Based Nutrition and Exercise for Sarcopenia Risk.
Acronym: S-TEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HSIAO MEI LAN (Other)
Responsible Party: Sponsor-Investigator, HSIAO MEI LAN, Master's Student and Geriatric Case Manager, Buddhist Tzu Chi General Hospital
Organization: Buddhist Tzu Chi General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB114-215-B; IRB114-215-B (Other: Research Ethics Committee Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Smart Technology; Nutrition and Exercise Intervention
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel arms: the Intervention Group (n=30) and the Control Group (n=30). Both groups will remain in their assigned arm for the entire 12-week study duration.
Masking Description: This study is an open-label randomized controlled trial (RCT) due to the complexity of the Line Bot intervention and the involvement of the same study personnel in both intervention delivery and data collection.
  Potential sources of bias are minimized through the following procedures:
  Random Allocation: Group assignment is conducted using sealed, opaque envelopes to ensure unbiased randomization.
  Objective Primary Outcomes: Primary outcomes such as muscle mass and physical function are assessed using standardized and quantifiable measurement instruments.
  Standardized Training: All study personnel responsible for data collection follow standardized operating procedures to ensure consistency across both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Technology-Assisted Exercise and Nutrition Program (Experimental): Participants in the intervention group (n=30) will receive a 12-week smart technology-assisted combined exercise and nutrition program. The intervention is delivered via a dedicated Line Bot platform, which provides: 1) Three progressive exercise training videos (resistance, aerobic, and balance) , **with the goal of participants completing five exercise sessions per week using the provided materials**. 2) Nutrition education videos focusing on protein intake. 3) Interactive features including daily reminders, protein intake calculation tools, and a digital diary with motivational elements to promote adherence and self-management.
  Interventions: Behavioral: The 12-week exercise component is delivered via the dedicated Line Bot platform. It includes three progressive exercise training videos (resistance, balance) . Participants are in
- Standard Outpatient Care (No Intervention): Participants in the control group (n=30) will receive standard outpatient care for sarcopenia risk management, which includes general health education pamphlets and regular follow-ups at the clinic. They will not receive any specialized exercise training, nutrition videos, or access to the Line Bot platform during the 12-week intervention period.

INTERVENTIONS:
Behavioral: The 12-week exercise component is delivered via the dedicated Line Bot platform. It includes three progressive exercise training videos (resistance, balance) . Participants are in — The 12-week progressive exercise program (resistance, aerobic, and balance training) is uniquely delivered and monitored via a dedicated **Line Bot platform**. This differentiates it from traditional in-person or non-interactive video programs. The platform includes interactive features like daily reminders and a digital diary to enhance adherence and support participant self-management, aiming for five exercise sessions per week.
  Arms: Smart Technology-Assisted Exercise and Nutrition Program

SUMMARY:
Sarcopenia, characterized by muscle loss and weakness, is a major health issue among older adults and impacts mobility and quality of life. This study addresses the current lack of long-term, technology-assisted support for managing this condition at home. This randomized controlled trial (RCT) will evaluate a 12-week smart-technology-based program for 60 older adults at risk of sarcopenia.

Intervention:

Participants in the intervention group will receive a technology-assisted program delivered through a Line Bot system. The platform provides personalized exercise training videos, nutrition education, daily reminders, and a point-based logging system to support adherence and monitor engagement. The control group will receive standard clinic-based care.

Purpose:

The study aims to examine whether the smart technology intervention can improve muscle mass, physical performance, quality of life, and self-management ability among older adults at risk of sarcopenia.

Expected Benefit:

The digital intervention is anticipated to offer a more effective, accessible, and sustainable approach compared with standard care, providing practical support for preventing muscle decline in community-dwelling older adults

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) is designed as a 12-week intervention to evaluate the efficacy of a smart technology-assisted nutrition and exercise program for community-dwelling older adults (aged ≥ 65 years) at risk of sarcopenia. Participants (N = 60) will be randomly assigned to either the intervention group (n = 30) or the control group (n = 30). Data will be collected at baseline, week 8 (mid-intervention), and week 12 (post-intervention).

Intervention Group:

Participants will receive the 12-week program delivered through a dedicated Line Bot platform. Core components include:

Exercise Training: Three progressive exercise videos (resistance, aerobic, and balance training) designed to enhance muscle function.

Nutrition Education: One video focusing on adequate protein intake and dietary habits essential for muscle maintenance.

Smart Technology Features: The Line Bot functions as a personalized case management tool, offering daily reminders for exercise and protein intake, an interactive calculator for estimating daily protein consumption, and a digital logging system with motivational rewards to support adherence and self-management behaviors.

Control Group:

Participants will receive standard outpatient care and general health education pamphlets. They will not receive access to the Line Bot system, exercise videos, or personalized support.

Primary outcome data will be collected at week 12. Statistical analyses will include descriptive statistics and inferential methods, such as repeated measures analysis of variance (ANOVA), to examine the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria

Score ≥ 11 on the SARC-CalF questionnaire, indicating risk of sarcopenia.

No evident functional impairment in the limbs and able to complete handgrip strength, walking speed, and muscle mass assessments.

Possesses basic reading, writing, and calculation abilities sufficient to understand study-related materials and complete informed consent and daily logs.

Owns a smartphone and has used it for at least one year, with basic operational ability (e.g., sending and receiving LINE messages, scanning QR codes).

Exclusion Criteria

Self-reported functional impairment in any limb.

Requires assistance from a wheelchair, walker, or cane for ambulation.

Has an implanted cardiac pacemaker.

Currently participating in, or planning to participate in, other physical training courses or nutrition programs during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Appendicular Skeletal Muscle Mass (ASM) by Bioelectrical Impedance Analysis (BIA) | Baseline (Week 0), Week 8, and Final Assessment at Week 12.
  The change in skeletal muscle mass will be assessed using Appendicular Skeletal Muscle Mass (ASM), derived from bioelectrical impedance analysis (BIA). The primary endpoint is the between-group difference in the absolute change in ASM (in kilograms) from baseline to the end of the 12-week intervention (Week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- BuddhistTCGH, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the lack of dedicated infrastructure and resources for data hosting, curation, and the formal management of external data access requests in this small, investigator-initiated study.